CLINICAL TRIAL: NCT04687449
Title: Curcumin in Management of Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial (C-COPD Trial)
Brief Title: Curcumin in Management of Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Danbury Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-1603
Record Dates: First submitted 2020-12-10; First posted 2020-12-29 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients with a diagnosis of COPD will be randomized to receive either a daily curcumin preparation or placebo for 90 days, in addition to the standard of care treatment.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Curcumin therapy added to standard COPD care (Active Comparator): Subjects will be given instructions to take 1 capsule twice daily for 90 days, 30 min before or 1 hour after meals, with a glass of water; if they develop upset stomach or diarrhea, then to take the medication with meals. This treatment will be in addition to the usual care that the hospital physician prescribe for them to treat the COPD.
  Interventions: Dietary Supplement: Curcumin therapy; Other: Standard care
- Active Comparator: Placebo with Standard COPD care (Active Comparator): Subjects will be given instructions to take 1 capsule twice daily for 90 days, 30 min before or 1 hour after meals, with a glass of water; if they develop upset stomach or diarrhea, then to take the medication with meals. This treatment will be in addition to the usual care that the hospital physician prescribe for them to treat the COPD.
  Interventions: Other: Placebo; Other: Standard care

INTERVENTIONS:
Dietary Supplement: Curcumin therapy — Clear capsules (made of vegetable cellulose) with turmeric extract (500 mg, 95% curcuminoids), Bioperine (5 mg, improves absorption), and inactive ingredients (microcrystalline cellulose, vegetable magnesium stearate, silicon dioxide).
  Arms: Active Comparator: Curcumin therapy added to standard COPD care
Other: Placebo — Clear capsules (made of vegetable cellulose) with inactive ingredients (lactose monohydrate and food color); the capsules will be matched in size and color of the content to the preparation used in the Curcumin capsule.
  Arms: Active Comparator: Placebo with Standard COPD care
Other: Standard care — The standard of care for COPD.

SUMMARY:
In this double-blind, placebo-controlled trial, 120 patients with a diagnosis of COPD will be randomized to receive either a daily curcumin preparation or placebo for 90 days, in addition to the standard of care treatment. The outcomes will be compared between the study arms. No dose escalation will be used.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) kills more than 3 million people worldwide every year. COPD is managed mainly by pharmacological therapy during the stable stage. Research illustrates many proven beneficial outcomes associated with the use of bronchodilators (beta-agonists and anticholinergics), inhaled and oral steroids to decrease the bronchial tree inflammation, some antibiotics, such as azithromycin, which have not only antibacterial but also some anti-inflammatory properties. However, these remedies have many limitations due to the development of adverse effects and resistance. Despite the treatment, symptoms related to COPD negatively affect patients' quality of life and limit their essential physical abilities, such as walking.

Although achievements have been made in the management of COPD, exacerbation (worsening or flare up) remains a leading cause for hospital admission. COPD exacerbation adversely affects patients' quality of and creates a significant financial burden on the healthcare system nationally and on a local level. Hospitals with excess readmission ratios for COPD are penalized financially by the Centers for Medicare and Medicaid Services. In Danbury Hospital, about 15% of patients admitted for COPD exacerbation are readmitted within 30 days on average.

Therefore, there is an urgent need for continued development of maintenance drugs for the treatment of COPD. Aside from the ordinary accepted pharmacological therapy approved for treatment of this chronic respiratory illness, some alternatives have pharmacologic properties that may potentially target the pathophysiologic processes involved in COPD.

Curcumin, a well-known polyphenol, is an active component of a plant Curcuma longa, commonly known as turmeric. Turmeric has been used for centuries as a spice and has recently become a widely used dietary supplement. Curcumin is reported to have anti-inflammatory properties by inhibiting NF-κB activation and IL-8,4,5 which are known to promote white blood cell activity and expression of COX-2 (enzyme responsible for production of inflammatory cytokines) involved in the pathophysiology of COPD. It has also been associated with the inhibition of cigarette smoke-induced NF-κB activation in bronchial epithelium in mice; in addition, it has been shown to revitalize steroid response in human cells.

The data on the effects of curcumin on inflammatory cytokines, as described above, has been derived from in vitro cell line and animal studies. While curcumin has been studied in humans for other inflammatory conditions (arthritis, gastrointestinal conditions, etc) to our knowledge, no human studies to explore its role in the management of COPD are available. As bronchial inflammation plays a key role in pathophysiology of COPD and curcumin has been shown to exhibit significant anti-inflammatory properties, we hypothesize that use of curcumin is associated with improvement in outcomes in patients with COPD.

Primary objective

1. To study if daily oral consumption of a curcumin preparation is associated with decreased health impairment in patients with COPD.

Secondary objectives

1. To study if daily oral consumption of a curcumin preparation is associated with improved functional exercise capacity among patients with COPD.
2. To study if daily oral consumption of a curcumin preparation is associated with decreased risk of an acute COPD exacerbation, and related hospital admission, in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form by the subject.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Clinical diagnosis of COPD, defined as having a smoking history of at least 10 pack-years, a ratio of post bronchodilator forced expiratory volume in 1 second [FEV1] to forced vital capacity of <70%, and a post bronchodilator FEV1 of <80% of the predicted value.
* Patient has not had an acute exacerbation of COPD for at least 4 weeks of time of screening.

Exclusion Criteria:

* Known allergic reactions to components of the study medication
* Use of turmeric as a spice or a dietary supplement within 3 months prior to enrollment
* Treatment with another investigational drug or other intervention at the time of enrollment
* Pregnancy or lactation
* Treatment with any chemotherapy agent, tacrolimus, talinolol, or sulfasalazine (due to the potential drug-drug interactions) at the time of enrolment
* Short-term steroid course received, for any reason, within 4 weeks prior to enrollment
* SGRQ-C is not available on the language preferred by the patient
* Patient is not able to undergo 6-minute walk due to a non-COPD related reason

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
St. George's Respiratory Questionnaire (SGRQ-C) score | Day 0 and 90
  Change in the 40-item version of the St. George's Respiratory Questionnaire (SGRQ-C) score: the score will be measured upon enrollment and at 90 days. It consists of 40 questions, and scored on 0 (no health impairment) to 100 (maximum health impairment) scale. The threshold for a clinically significant difference between groups of patients and for changes within groups of patients is four units.

SECONDARY OUTCOMES:
Performance on the 6-minute walk test (6MWT) | Day 0 and 90
  Change in the 6-minute walk test (6MWT) result (in meters): the test will be administered upon enrollment and at 90 days.
Time to the first acute exacerbation of COPD | 6 months
  Difference in the time from initiation of the study medication to the first acute COPD exacerbation. Participants will be contacted over the phone 6 months after taking the first dose of the study medication, to inquire about outpatient and inpatient encounters for acute worsening of COPD occurred after the 90-day follow-up appointment; the participants' medical records will also be reviewed to determine if the reported encounters occurred due to acute COPD exacerbation as diagnosed by a medical provider and also to determine if COPD exacerbation occurred in those participants who could not be reached over the phone.
Relative risk of the acute COPD exacerbation | 6 months
  Relative risk of the acute COPD exacerbation occurred during the study will be analyzed descriptively by calculating average occurrence (number of incidences in population over the 6-month period) in both study groups. Participants will be contacted over the phone 6 months after taking the first dose of the study medication, to inquire about outpatient and inpatient encounters for acute worsening of COPD occurred after the 90-day follow-up appointment; the participants' medical records will also be reviewed to determine if the reported encounters occurred due to acute COPD exacerbation as diagnosed by a medical provider and also to determine if COPD exacerbation occurred in those participants who could not be reached over the phone.
Relative risk of hospital admission for acute COPD exacerbation. | 6 months
  Relative risk of hospital admission for acute COPD exacerbation occurred during the study will be analyzed descriptively by calculating average occurrence (number of incidences in population over the 6-month period) in both study groups. Participants will be contacted over the phone 6 months after taking the first dose of the study medication, to inquire about outpatient and inpatient encounters for acute worsening of COPD occurred after the 90-day follow-up appointment; the participants' medical records will also be reviewed to determine if the reported encounters occurred due to acute COPD exacerbation as diagnosed by a medical provider and also to determine if COPD exacerbation occurred in those participants who could not be reached over the phone.

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Sostin, MD, Principal Investigator — Danbury Hospital, Nuvance Health
Locations (1):
- Pulmonary and Sleep Medicine clinic, Danbury, Connecticut, United States

REFERENCES:
- [Background] Rabe KF, Watz H. Chronic obstructive pulmonary disease. Lancet. 2017 May 13;389(10082):1931-1940. doi: 10.1016/S0140-6736(17)31222-9. Epub 2017 May 11. PMID 28513453
- [Background] Miravitlles M, Ribera A. Understanding the impact of symptoms on the burden of COPD. Respir Res. 2017 Apr 21;18(1):67. doi: 10.1186/s12931-017-0548-3. PMID 28431503
- [Background] Shah T, Churpek MM, Coca Perraillon M, Konetzka RT. Understanding why patients with COPD get readmitted: a large national study to delineate the Medicare population for the readmissions penalty expansion. Chest. 2015 May;147(5):1219-1226. doi: 10.1378/chest.14-2181. PMID 25539483
- [Background] Shishodia S, Potdar P, Gairola CG, Aggarwal BB. Curcumin (diferuloylmethane) down-regulates cigarette smoke-induced NF-kappaB activation through inhibition of IkappaBalpha kinase in human lung epithelial cells: correlation with suppression of COX-2, MMP-9 and cyclin D1. Carcinogenesis. 2003 Jul;24(7):1269-79. doi: 10.1093/carcin/bgg078. Epub 2003 May 9. PMID 12807725
- [Background] Yuan J, Liu R, Ma Y, Zhang Z, Xie Z. Curcumin Attenuates Airway Inflammation and Airway Remolding by Inhibiting NF-kappaB Signaling and COX-2 in Cigarette Smoke-Induced COPD Mice. Inflammation. 2018 Oct;41(5):1804-1814. doi: 10.1007/s10753-018-0823-6. PMID 29961171
- [Background] Suzuki M, Betsuyaku T, Ito Y, Nagai K, Odajima N, Moriyama C, Nasuhara Y, Nishimura M. Curcumin attenuates elastase- and cigarette smoke-induced pulmonary emphysema in mice. Am J Physiol Lung Cell Mol Physiol. 2009 Apr;296(4):L614-23. doi: 10.1152/ajplung.90443.2008. Epub 2009 Jan 23. PMID 19168576
- [Background] Zhang M, Xie Y, Yan R, Shan H, Tang J, Cai Y, Yin J, Chen M, Zhang J, Yang X, Zhang Q, Li Y. Curcumin ameliorates alveolar epithelial injury in a rat model of chronic obstructive pulmonary disease. Life Sci. 2016 Nov 1;164:1-8. doi: 10.1016/j.lfs.2016.09.001. Epub 2016 Sep 4. PMID 27600540
- [Background] Vecchi Brumatti L, Marcuzzi A, Tricarico PM, Zanin V, Girardelli M, Bianco AM. Curcumin and inflammatory bowel disease: potential and limits of innovative treatments. Molecules. 2014 Dec 16;19(12):21127-53. doi: 10.3390/molecules191221127. PMID 25521115
- [Background] Daily JW, Yang M, Park S. Efficacy of Turmeric Extracts and Curcumin for Alleviating the Symptoms of Joint Arthritis: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. J Med Food. 2016 Aug;19(8):717-29. doi: 10.1089/jmf.2016.3705. PMID 27533649
- [Background] Jones PW. Interpreting thresholds for a clinically significant change in health status in asthma and COPD. Eur Respir J. 2002 Mar;19(3):398-404. doi: 10.1183/09031936.02.00063702. PMID 11936514
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Solway S, Brooks D, Lacasse Y, Thomas S. A qualitative systematic overview of the measurement properties of functional walk tests used in the cardiorespiratory domain. Chest. 2001 Jan;119(1):256-70. doi: 10.1378/chest.119.1.256. PMID 11157613
- [Background] Singh D, Agusti A, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Criner GJ, Frith P, Halpin DMG, Han M, Lopez Varela MV, Martinez F, Montes de Oca M, Papi A, Pavord ID, Roche N, Sin DD, Stockley R, Vestbo J, Wedzicha JA, Vogelmeier C. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease: the GOLD science committee report 2019. Eur Respir J. 2019 May 18;53(5):1900164. doi: 10.1183/13993003.00164-2019. Print 2019 May. PMID 30846476
- [Background] Rennard S, Thomashow B, Crapo J, Yawn B, McIvor A, Cerreta S, Walsh J, Mannino D. Introducing the COPD Foundation Guide for Diagnosis and Management of COPD, recommendations of the COPD Foundation. COPD. 2013 Jun;10(3):378-89. doi: 10.3109/15412555.2013.801309. PMID 23713598
- [Background] Fung FY, Wong WH, Ang SK, Koh HL, Kun MC, Lee LH, Li X, Ng HJ, Tan CW, Zhao Y, Linn YC. A randomized, double-blind, placebo- controlled study on the anti-haemostatic effects of Curcuma longa, Angelica sinensis and Panax ginseng. Phytomedicine. 2017 Aug 15;32:88-96. doi: 10.1016/j.phymed.2017.04.004. Epub 2017 Apr 10. PMID 28732813
- [Background] Liu AC, Zhao LX, Lou HX. Curcumin alters the pharmacokinetics of warfarin and clopidogrel in Wistar rats but has no effect on anticoagulation or antiplatelet aggregation. Planta Med. 2013 Jul;79(11):971-7. doi: 10.1055/s-0032-1328652. Epub 2013 Jun 27. PMID 23807811